CLINICAL TRIAL: NCT01560390
Title: Use of Ketamine Associate With an Opioid for Sedation in ICU : a Randomized Controlled Double Blind Study
Brief Title: Use of Ketamine Associate With an Opioid for Sedation in ICU
Acronym: KetaRea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0108
Record Dates: First submitted 2011-11-17; First posted 2012-03-22 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Sedation for Mechanical Ventilation
Keywords: Sedation; ICU; Ketamine; Confusion; Hyperalgesia
MeSH Terms: conditions — Confusion; Hyperalgesia | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Rémifentanil + Kétamine (Other): to evaluate the impact of ketamine associated to an opioid for sedation of mechanically ventilated critically ill patients versus placebo. Sedation will be drive by nurses according to an algorithm. The investigators will evaluate the quantity of opioates used in each arm and the safety of ketamine.
  Interventions: Drug: Rémifentamil + KETAMINE; Drug: ketamine
- Rémifentanil + Placebo (Other): to evaluate the impact of ketamine associated to an opioid for sedation of mechanically ventilated critically ill patients versus placebo. Sedation will be drive by nurses according to an algorithm. The investigators will evaluate the quantity of opioates used in each arm and the safety of ketamine.
  Interventions: Drug: Rémifentamil + KETAMINE; Drug: ketamine

INTERVENTIONS:
Drug: Rémifentamil + KETAMINE — All consecutive mechanically ventilated patients admitted in the ICU will be randomized to receive an infusion of 0.15 mg/kg/h of kétamine or placebo. Nurses and physicians will be blinded of the allocation arm. The infusion of ketamine will be stopped as soon as remifentanil will be discontinued by the physician.
Drug: ketamine — to evaluate the impact of ketamine associated to an opioid for sedation of mechanically ventilated critically ill patients versus placebo. Sedation will be drive by nurses according to an algorithm. The investigators will evaluate the quantity of opioates used in each arm and the safety of ketamine.

SUMMARY:
The aim of the study is to evaluate the impact of ketamine associated to an opioid for sedation of mechanically ventilated critically ill patients versus placebo. Sedation will be drive by nurses according to an algorithm. The investigators will evaluate the quantity of opioates used in each arm and the safety of ketamine.

DETAILED DESCRIPTION:
All consecutive mechanically ventilated patients admitted in the intensive care unit (ICU)will be randomized to receive an infusion of 0.15 mg/kg/h of kétamine or placebo. Nurses and physicians will be blinded of the allocation arm. The infusion of ketamine will be stopped as soon as remifentanil will be discontinued by the physician.

ELIGIBILITY:
Inclusion Criteria:

* all patients under mechanical ventilation

Exclusion Criteria:

* pregnant
* psychotic
* chronic use of opiates
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2011-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Amount of opiate used between study enrollment and mechanical ventilation withdrawal. | after 24 hours

SECONDARY OUTCOMES:
Confusion Duration assessed by CAM-ICU | after 24 hours
mechanical ventilation duration | after 24 hours
ICU length of stay | after 24 hours
Mortality at D28 | at day 28
hyperalgesia during sedation | after 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel CONSTANTIN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France